CLINICAL TRIAL: NCT04674501
Title: A Prospective Cohort Study of Patients Receiving Radiotherapy for Thoracic and Breast Cancer and the Related Cardiotoxicity Following Treatment (RACCOON)
Brief Title: Radiotherapy for Thoracic and Breast Cancer and the Related Cardiotoxicity Following Treatment (RACCOON)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2020-1093
Record Dates: First submitted 2020-12-04; First posted 2020-12-19 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Patients Who Receive Thoracic Irradiation
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Thoracic irradiation: A cohort of cancer patients who receive thoracic irradiation. Patients with any type of malignancy, such as lung cancer, breast cancer, esophageal cancer, or thymoma, are eligible as long as the patients undergo thoracic irradiation.
  Interventions: Procedure: Cardiac evaluation and blood sampling

INTERVENTIONS:
Procedure: Cardiac evaluation and blood sampling — Patients in this cohort will undergo cardiac evaluation before and after thoracic irradiation.
  The dose-volume parameters for each cardiac substructures will be estimated using artificial intelligence-based auto-segmentation of the heart in CT images. Dose-volume parameters that predict cardiotoxicity will be analyzed.
  The patients who developed cardiotoxicity will undergo blood sampling to establish cardiomyocytes derived from induced pluripotent stem cells, which will be used for identifying the mechanisms of radiation-induced cardiotoxicity and therapeutic targets.

SUMMARY:
The purpose of this study is to investigate the risk factors and mechanisms of cardiotoxicity following thoracic radiotherapy and to provide insights in preventing radiation-related cardiotoxicity.

-Condition or disease : Thoracic irradiation -Intervention/treatment : Cardiac evaluation, Blood sampling

DETAILED DESCRIPTION:
Cancer patients who undergo thoracic irradiation receive a certain amount of dose to the heart. Cardiotoxicity may occur in some patients several years after radiotherapy due to the late effect of radiation. Considering that cardiotoxicity is often lethal, screening and preventing radiation-induced cardiotoxicity is crucial in patients receiving thoracic irradiation.

Patients in this cohort will undergo cardiac evaluation before and after thoracic irradiation. The dose-volume parameters for each cardiac substructures will be estimated using artificial intelligence-based auto-segmentation of the heart in CT images. Dose-volume parameters that predict cardiotoxicity will be analyzed. Among the patients who developed cardiotoxicity, blood sampling will be performed to establish cardiomyocytes derived from induced pluripotent stem cells, which will be used for identifying the mechanisms of radiation-induced cardiotoxicity and therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with solid cancer who are subject to thoracic irradiation.
2. Patients who are 20 years old or older
3. Eastern Cooperative Oncology Group Performance Status Scale 0-2
4. Patients with cognitive abilities to receive virtual reality information

Exclusion Criteria:

1. Patients with a history of previous thoracic irradiation
2. Patients who refused consent
3. Patients with a history of heart failure before radiotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with solid tumors who receive thoracic irradiation
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Cardiotoxicity rate | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years
Cancer-specific survival | 2 years
Progression-free survival | 2 years
Other toxicity rates | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Hong In Yoon, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei Cancer Center, Yonsei University College of Medicine, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No